CLINICAL TRIAL: NCT03206151
Title: Open, Randomized, Controlled, Multicenter Phase III Study Comparing CMAB009 Plus FOLFIRI Versus FOLFIRI Alone as First-line Treatment for Epidermal Growth Factor Receptor-expressing, RAS/BRAF Wild-type, Metastatic Colorectal Cancer
Brief Title: CMAB009 Combined With FOLFIRI First-line Treatment in Patients With RAS/BRAF Wild-type, Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 009mCRCIIIP
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — CMAB009; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMAB009 + FOLFIRI (Experimental): Drug: CMAB009(recombinant chimeric anti-EGFR monoclonal antibody injection), will be administered every 7 days at an initial dose of 400mg/m^2 and 250mg/m^2 for subsequent infusions until progression of disease , withdrawal of consent, or unacceptable toxicity.
  Drug: Irinotecan bi-weekly irinotecan infusion of 180mg/m^2 on Day 1. Drug: Folinic Acid infusion 400mg/m^2 of folinic acid in on Day 1. Drug: 5-Fluorouracil bolus 5-Fluorouracil bolus of 400mg/m^2 followed by a 46-48 h continuous infusion of 2400mg/m^2.
  every 2 weeks until progression of disease , withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: CMAB009; Drug: Irinotecan; Drug: Folinic acid; Drug: 5-fluorouracil
- FOLFIRI (Active Comparator): FOLFIRI Drug: Irinotecan bi-weekly irinotecan infusion of 180mg/m^2 on Day 1. Drug: Folinic Acid infusion 400mg/m^2 of folinic acid in on Day 1. Drug: 5-Fluorouracil bolus 5-Fluorouracil bolus of 400mg/m^2 followed by a 46-48 h continuous infusion of 2400mg/m^2.
  every 2 weeks until progression of disease , withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: Irinotecan; Drug: Folinic acid; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: CMAB009 — for injection only
  Other Names: Eribitux
  Arms: CMAB009 + FOLFIRI
Drug: Irinotecan — for injection only
  Other Names: Camptosar
Drug: Folinic acid — for injection only
  Other Names: leucovorin
Drug: 5-fluorouracil — for injection only
  Other Names: Fluoroplex

SUMMARY:
Drugs used against cancer work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as CMAB009, can block tumor growth in different ways. Giving combination chemotherapy together with CMAB009 as first treatment after diagnosis of a metastatic colorectal cancer（first-line treatment）may improve the treatment efficacy. However, it is not yet known whether giving combination chemotherapy together with CMAB009 is more effective than combination chemotherapy alone. This open-label trial investigates the effectiveness of CMAB009 in combination with a standard and effective chemotherapy FOLFIRI（5-Fluorouracil /Folinic acid plus Irinotecan）for RAS/BRAF wild-type, metastatic colorectal cancer in first-line setting, compared to the same chemotherapy alone.

DETAILED DESCRIPTION:
Patients will be randomly assign in one of the two groups to either receive the combination chemotherapy alone or with CMAB009 and will then be treated until progression of the disease or unacceptable toxicity occurred. Regular efficacy assessments（every 8 weeks）based on imaging will be performed throughout the study together with regular safety assessments.

After participant discontinuation from the trial, regular updates on further treatments and survival status will be requested from the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, Aged ≥18 years and ≤75 years
2. Diagnosis of histologically confirmed adenocarcinoma of the colon or rectum
3. First occurrence of metastatic disease(not curatively resected)
4. RAS/BRAF wild-type status in tumor tissue
5. At least one measurable lesion by computer tomography(CT) or magnetic resonance imaging (MRI)according to RECIST1.1 criteria (not in an irradiated area)
6. Eastern Cooperative Oncology Group(ECOG)performance status of 0 or 1 at trial entry
7. Life expectancy of at least 3 months
8. Medically accepted effective contraception if procreative potential exists(applicable for both male and female subjects until at least 90 days after the last dose of trial treatment)
9. Recovery from relevant toxicity due to previous treatment before trial entry
10. Signed the informed consent form voluntarily

Exclusion Criteria:

1. Radiotherapy or surgery（excluding prior diagnostic biopsy）in the 30 days before trial treatment
2. Hepatic, marrow, liver and renal function as follows:

   Marrow: white blood cell count <3.0 × 109/L with neutrophils<1.5 × 109/L, platelet count<100×109/L and hemoglobin<90 g/L; Liver function: Total bilirubin >1.5 × upper limit of reference range; Aspartate transaminase (AST) and alanine transaminase (ALT) > 2.5 × upper limit of reference range , or> 5 × upper reference range in subjects with liver metastasis; Renal function: Serum creatinine >1.5 × upper limit of reference range, or creatinine clearance<50 mL/min
3. Previous chemotherapy for CRC adjuvant treatment if terminated <12 months before diagnosis of recurrence or metastatic disease
4. Previous treatment with anti-EGFR monoclonal antibody, epidermal growth factor receptor tyrosine kinase inhibitor, or other EGFR targeted inhibitors(such as cetuximab, Nimotuzumab, or panitumumab)
5. Known hypersensitivity or allergic reactions against any of the components of the trial treatments
6. History of organ allograft, autologous stem cell transplantation, or allogeneic stem cell transplantation
7. Other non-permitted concomitant anti-cancer therapies
8. Known brain metastasis and/or leptomeningeal disease
9. Previous malignancy other than CRC in the last 5 years except basal cell cancer of the skin or preinvasive cancer of the cervix
10. Participation in another clinical trial within the past 30 days
11. Concurrent chronic systemic immune therapy or hormone therapy except physiologic replacement
12. Any unstable systemic disease, such as active infection, uncontrolled hypertension, unstable angina pectoris, angina in the last 3 months, cardiac failure of New York Heart Association classes ≥II, history of myocardial infarction, serious cardiac arrhythmias that require drug treatment, liver, kidney or metabolic disease in the last 6 months
13. Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
14. severe bone marrow function failure
15. Any disease, metabolic disorders, or physical/laboratory examination suspected, or patients with high risk of complications
16. Known and declared history of human immunodeficiency virus(HIV)infection
17. HBV-DNA >1.0 × 103copy
18. Pregnancy or breastfeeding
19. Alcohol or drug abuse
20. Legal incapacity or limited legal capacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Tumor assessments are conducted every 8 weeks after randomization until the end of the study, an average of 1 year.
  The PFS duration (in months) is determined by a specially authorized Independent Radiology Review Committee (IRaC) through blinded review of imaging data. It is defined as the time from randomization to the first confirmed progression of disease by imaging or death from any cause within 90 days after the last tumor assessment or randomization, whichever is later (equivalent to 1.5 times the interval between two consecutive tumor assessments).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Tumor assessments are conducted every 8 weeks after randomization until the end of the study, an average of 1 year.
  The objective response rate is calculated as the percentage of evaluable subjects with complete response (CR) and partial response (PR) (ORR = CR + PR).
Overall Survival（OS） | From randomization until the end of the study, an average of 1 year.
  Defined as the time from randomization to death (in months). For subjects still alive or lost to follow-up as of the data analysis cutoff date, survival is censored at the subject's last known alive time.
Disease Control Rate (DCR) | Tumor assessments are conducted every 8 weeks after randomization until the end of the study, an average of 1 year.
  Refers to the percentage of subjects with the best response of complete response (CR), partial response (PR), and stable disease (SD) according to RECIST 1.1 criteria (DCR = CR + PR + SD).
Time to Response (TTR) | Tumor assessments are conducted every 8 weeks after randomization until the end of the study, an average of 1 year.
  For subjects with the best response of CR or PR according to RECIST 1.1 criteria, the time from randomization to the first occurrence of response (CR or PR) according to RECIST 1.1.
Quality of Life Assessment Indicators | Assessments are conducted at baseline and subsequent visits every 8 weeks until withdrawal from the study and entry into the follow-up period.
  Quality of life assessment (QOL) is conducted using the EORTC QLQ-C30 questionnaire, with individual item categorical scores linearly transformed to a 0-100 scale.
Resection Rate of Hepatic Metastasis | From randomization to the end of study
  The resection rate of hepatic metastasis is calculated as the number of subjects achieving complete resection (R0 resection) divided by the total number of subjects.
Safety Endpoint | From enrollment to the end of study
  Drug exposure, All types of AEs and incidence rates, Mortality rate and causes of death, Safety laboratory tests, Vital signs and Immunogenicity.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi Professor, Ph.D, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Yi Ba Professor, Ph.D, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (2):
- China (2):
  - Cancer hospital Chinese academy of medical sciences, Beijing, Beijing Municipality
  - Tianjing medical university cancer institute and hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shi Y, Ba Y, Wang J, Xiong J, Gu K, Chen Y, Zheng Z, Wang Z, Guo W, Cheng Y, Yin X, Liu Y, Bai Y, Li E, Li Q, Zhu L, Li W, Jiang D, He J, Chen J, Sun J, Hou S. First-line treatment of anti-EGFR monoclonal antibody cetuximab beta plus FOLFIRI versus FOLFIRI alone in Chinese patients with RAS/BRAF wild-type metastatic colorectal cancer: a randomized, phase 3 trial. Signal Transduct Target Ther. 2025 May 7;10(1):147. doi: 10.1038/s41392-025-02229-4. PMID 40328753